CLINICAL TRIAL: NCT00873236
Title: Dynamic Contrast Enhanced MRI (DCE-MRI) Assessment of the Vascular Changes Induced With Bevacizumab Alone and in Combination With Interferon-α in Patients With Advanced Renal Cell Carcinoma
Brief Title: MRI Scans of Blood Vessel Changes Caused by Bevacizumab Alone or Given Together With Interferon Alpha-2a in Treating Patients With Stage III or Stage IV Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Vernon Cancer Centre at Mount Vernon Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Diagnostic
Other Study IDs: MTVERNHOSP-RD2007-114; CDR0000637812 (Registry Identifier: PDQ (Physician Data Query)); ENH-RD2007-114; EUDRACT-2008-006414-19; EU-20917
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-03

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Bevacizumab; Interferon alpha-2

ARMS (3):
- Arm I (Experimental): Patients receive bevacizumab IV over 30-90 minutes once every 2 weeks.
  Interventions: Biological: bevacizumab
- Arm II (Experimental): Patients receive bevacizumab as in arm I and low-dose recombinant interferon alpha-2a subcutaneously (SC) 3 times weekly beginning on day 0.
  Interventions: Biological: bevacizumab; Biological: recombinant interferon alpha-2a
- Arm III (Experimental): Patients receive bevacizumab as in arm I and standard-dose recombinant interferon alpha-2a SC 3 times weekly beginning on day 0.
  Interventions: Biological: bevacizumab; Biological: recombinant interferon alpha-2a

INTERVENTIONS:
Biological: bevacizumab — Given IV
Biological: recombinant interferon alpha-2a — Given SC
  Arms: Arm II; Arm III

SUMMARY:
RATIONALE: Comparing results of MRI scans done after bevacizumab may help doctors predict a patient's response to treatment and help plan the best treatment. It is not yet known whether giving bevacizumab alone is more effective than giving bevacizumab together with interferon alpha-2a in detecting kidney cancer.

PURPOSE: This randomized phase II trial is studying MRI scans of blood vessel changes caused by bevacizumab to see how well it works compared with bevacizumab given together with interferon alpha-2a in treating patients with stage III or stage IV kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish whether bevacizumab-induced changes in dynamic contrast-enhanced (DCE)-MRI vascular parameters are significantly enhanced by recombinant interferon alpha-2a.
* To establish whether there is an interferon alpha-2a dose response in potentiating bevacizumab-induced changes in DCE-MRI vascular parameters.

Secondary

* To correlate changes in DCE-MRI vascular parameters for each treatment group with progression-free survival.
* To correlate changes in DCE-MRI vascular parameters for each treatment group with tumor response and changes in tumor size.
* To correlate changes in DCE-MRI vascular parameters for each treatment group with other surrogate biomarkers.
* To assess the degree of change in baseline K^trans within each arm of treatment.
* To investigate changes in diffusion and blood oxygen-level dependent MRI and their correlation with other pharmacodynamic endpoints.
* To assess the efficacy and safety profile of bevacizumab monotherapy or in combination with low or standard doses of recombinant interferon alpha-2a.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive bevacizumab IV over 30-90 minutes once every 2 weeks.
* Arm II: Patients receive bevacizumab as in arm I and low-dose recombinant interferon alpha-2a subcutaneously (SC) 3 times weekly beginning on day 0.
* Arm III: Patients receive bevacizumab as in arm I and standard-dose recombinant interferon alpha-2a SC 3 times weekly beginning on day 0.

After 8 weeks of treatment, recombinant interferon alpha-2a dosage may be modified or discontinued at the discretion of the investigator. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients undergo dynamic contrast-enhanced (gadopentetate dimeglumine) MRI scans at baseline and weeks 2 and 6. Peripheral blood and serum samples are collected at baseline and weeks 2, 6, and 8 for analysis of surrogate biomarkers by flow cytometry and mRNA analysis by PCR. Archival histopathological specimens are analyzed by IHC, fluorescence resonance-energy transfer, and fluorescence lifetime-imaging. Urine samples are also collected at baseline for proteomic profiling by MALDI-TOF.

After completion of study treatment, patients are followed at 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced renal cell carcinoma

  * Metastatic (stage IV) disease
  * Locally advanced (unresectable stage III) disease
* Previously untreated disease
* Majority component of conventional clear-cell type is mandatory (tumors of mixed histology should be categorized by the predominant cell type)
* Good- or intermediate-prognosis disease as defined by Motzer score
* Lesions measurable by RECIST criteria and amenable to dynamic contrast-enhanced MRI scanning
* No brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8 g/dL (may be transfused to maintain or exceed this level)
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT < 2.5 times ULN (< 5 times ULN in patients with liver metastases)
* Serum creatinine ≤ 1.5 times ULN
* Urine dipstick for proteinuria < 2+ OR < 1 g of protein in 24-hour urine collection
* INR ≤ 1.5
* Not pregnant or nursing
* Negative pregnancy test
* Fertile women must use effective contraception during and for 9 months after completion of study treatment
* No significant cardiovascular disease, defined as any of the following, within the past 6 months:

  * NYHA class II-IV congestive heart failure
  * Unstable angina pectoris
  * Myocardial infarction
* No significant vascular disease (e.g., aortic aneurysm, aortic dissection) or symptomatic peripheral vacular disease
* No evidence or history of recurrent thromboembolism (> 1 episode of deep venous thrombosis/pulmonary embolism) within the past 6 months, bleeding diathesis, or coagulopathy
* No inadequately controlled hypertension (defined as a BP of > 150 mm Hg systolic and/or > 100 mm Hg diastolic on medication)
* No history of hypertensive crisis or hypertensive encephalopathy
* No stroke or transient ischemic attack within the past 6 months
* No abdominal or tracheoesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No HIV or hepatitis B or C infection
* No active clinically serious bacterial or fungal infections (> CTCAE grade 2)
* No other infection > CTCAE grade 2
* No concurrent active second malignancy within the past 3 years other than nonmelanoma skin cancers or post-treatment for localized prostate cancer
* No gross ascites
* No seizure disorder requiring medication
* No serious non-healing wound, ulcer, or bone fracture
* No contraindications to MRI scanning (e.g., history of claustrophobia or metal fragment implantation)
* No history of allergic reactions to contrast agents
* No other significant medical illness or medically significant abnormal laboratory finding that would, in the investigator's opinion, make the patient inappropriate for this study, or would increase the risk associated with the patient's participation in the study

PRIOR CONCURRENT THERAPY:

* More than 28 days since prior major surgery (including open biopsy) or radiotherapy and recovered
* More than 14 days since prior palliative radiotherapy to painful bone lesions and recovered

  * Concurrent palliative radiotherapy for local pain control allowed
* More than 7 days since prior core biopsy or other minor surgical procedure, excluding placement of a vascular access device
* More than 30 days since prior and no other concurrent investigational agents
* No concurrent chronic daily intake of aspirin ≥ 325 mg/day or clopidogrel > 75 mg/day, or steroids (prednisone > 12.5 mg/day or dexamethasone > 2 mg/day), excluding inhaled steroids
* No concurrent bone marrow transplantation or stem cell rescue
* Concurrent anticoagulation allowed provided INR < 3 and INR is therapeutic on a stable dose of coumarin-type anticoagulation or if patient is on a stable dose of low molecular weight heparin for > 2 weeks at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-04

PRIMARY OUTCOMES:
Dynamic contrast-enhanced MRI defined changes in K-trans after 6 weeks of bevacizumab monotherapy or bevacizumab and low- or standard-dose recombinant interferon alpha-2a

SECONDARY OUTCOMES:
Change in vascular permeability (K-trans) and tumor hypoxia at 2 and 6 weeks post-commencement of treatment
Best overall response
Progression-free survival
Time to progression
Treatment duration of bevacizumab and recombinant interferon alpha-2a
Treatment withdrawal
Dose modification
Incidence of adverse events
Number of circulating endothelial cells, circulating endothelial progenitors, and proangiogenic monocytic cells
Angiogenic factors (e.g., VEGF) and hypoxia-regulated markers
Correlation of DCE-MRI defined changes in K-trans with clinical response
Correlation of DCE-MRI defined changes in K-trans with surrogate biomarkers
Analysis of diffusion MRI and blood oxygen-level dependent MRI changes and comparison with other pharmacodynamic markers

CONTACTS AND LOCATIONS:
Overall Officials: Paul Nathan, MD, Principal Investigator — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (5):
- United Kingdom (5):
  - Addenbrooke's Hospital, Cambridge, England
  - Royal Marsden - London, London, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Churchill Hospital, Oxford, England
  - Royal Marsden - Surrey, Sutton, England